CLINICAL TRIAL: NCT01842490
Title: Can Serum Biomarker of Plaque Vulnerability be Identified Through the Contrast-enhanced Ultrasound of Carotid Artery
Brief Title: Serum Biomarker of Plaque Vulnerability and Contrast Ultrasound of Carotid Artery
Status: Completed | Type: Observational
Sponsor: Kyunghee University Medical Center (Other)
Responsible Party: Principal Investigator, Weon Kim, Assoiciate Professor, Kyunghee University Medical Center
Other Study IDs: INCA
Record Dates: First submitted 2013-03-23; First posted 2013-04-29 (Estimated); Last update posted 2014-08-25 (Estimated); Status verified 2013-04

CONDITIONS: Intraplaque Neovascularization Evaluated by Carotid Enhanced Ultrasound Well Reflect the Plaque Vulnerability
Keywords: Biomarker; Carotid enhanced ultrasound; Intraplaque neovascularization

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: Yes

SUMMARY:
No serum biomarker has qualified for clinical use until now. However several biomarkers, especially markers of inflammatory or proteolytic activity seem to promising in the identification of vulnerable plaques. Moreover, recent study confirmed that contrast-enhanced ultrasound imaging(CEUS) can visualize intraplaque neovascularization and represent the plaque vulnerability. In this study we try to identify indicators through analysis of the relationship between plaque neovascularization seen by CEUS and well known biomarkers such as serum matrix metalloproteinase(MMP)-2, MMP-9, cathepsin family(L,S,V), cystatin C, lipoprotein phospholipase A2, and hs-crp

ELIGIBILITY:
Inclusion Criteria:

* patients with carotid plaques size more than 2mm by carotid ultrasound

Exclusion Criteria:

* known allergy to albumin, or to the ultrasound contrast agent
* the patients with history of carotid endarterectomy and carotid stent
* acute myocardial infarction, cardiogenic shock
* connective tissue disease and malignancy
* creatinine clearance lower than 30ml/min and the history of dialysis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The patients were selected from those who admitted due to chest pain and underwent carotid duplex ultrasound examination at KyungHee university medical center, Seoul, South Korea.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2010-05; Primary Completion 2013-10 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Peak plasma concentration of Biomarker that is statistically significant different according to the presence of intraplaque neovascularization on contrast enhanced ultrasound of carotid artery | after performing contrast enhanced ultrasound of carotid artery, upto 3 hospital days

SECONDARY OUTCOMES:
the number of the patients with history of cardiovascular event including myocardial infarction, cerebral vascular event and peripheral arterial disease and the number of 1 year clinical outcome of cardiovascular event | after performing contrast enhanced ultrasound of carotid artery, upto 1 year clinical follow up

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Cardiology, Department of Internal Medicine, Kyung Hee University School of Medicine, Seoul, Seoul, South Korea